CLINICAL TRIAL: NCT04895800
Title: An Evaluation of the Effects of a Non-Caffeinated Energy Die-tary Supplement on Cognitive and Physical Performance: A Randomized Double-Blind Placebo-Controlled Study
Brief Title: An Evaluation of the Effects of a Non-Caffeinated Energy Dietary Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Jaime Tartar, Professor, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-563
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: A Randomized Double-Blind Placebo-Controlled Study
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Herbal Supplement (Experimental): (Phytovive™); comprised of Bacopa monnieri bacosides, Kaempferia parviflora methoxy flavones, pomegranate peel polyphenols, and Moringa oleifera leaf saponins)
  Interventions: Dietary Supplement: Phytovive
- Caffeine (Active Comparator): Green tea caffeine extract (170 mg; to deliver 34 mg caffeine [20% natural caffeine]),
  Interventions: Dietary Supplement: Caffeine
- Placebo (Placebo Comparator): Flavored placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phytovive — Bacopa monnieri bacosides, Kaempferia parviflora methoxy flavones, pomegranate peel polyphenols, and Moringa oleifera leaf saponins)
  Arms: Herbal Supplement
Dietary Supplement: Placebo — Natural Flavors [Chocolate, Caramel, Vanilla Cream], Silica, Inulin, Sucralose)
  Arms: Placebo
Dietary Supplement: Caffeine — Caffeine (Green tea caffeine extract (170 mg; to deliver 34 mg caffeine [20% natural caf-feine])
  Arms: Caffeine

SUMMARY:
This study tested the effects of a botanical blend to a caffeine and a placebo condition on 1) self-reported alertness, anxiety, and headaches 2) multiple measures of attention 3) physical performance and 4) stress biomarkers.

DETAILED DESCRIPTION:
This study aimed to build on this work by investigating the possibility that a specific botanical blend (Phytovive™); comprised of Bacopa monnieri bacosides, Kaempferia parviflora methoxy flavones, pomegranate peel polyphenols, and Moringa oleifera leaf saponins) could improve cognitive and physical performance. To this end, this study was a randomized, double-blind, placebo-controlled 21-day parallel study on 36 healthy adults. The study compared the effects of the botanical blend at baseline to a caffeine and a placebo condition on 1) self-reported alertness, anxiety, and headaches 2) multiple measures of attention 3) physical performance and 4) stress biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females from 18 to 50 years (inclusive) of age who are physically active and have been engaging in athletic and sporting endeavors consistently over a period of 6 months at minimum
* BMI 18.0 (normal) to 34.9 (obese, class I) kg/ m2 inclusive
* Agrees to maintain a stable lifestyle with no change in exercise or diet for the duration of the study
* Current consumer of caffeine either through caffeinated beverages or foods
* Non-smoker
* Able to physically exercise, to run on a treadmill at moderate to high intensity for a brief time (typically less than 20 min)
* Participants with normal blood pressure or participants with hypertension that is controlled (BP < 160/90 and who are on medication at a stable dose (same dose for ≥90 days)
* Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, carry out all study-related procedures, communicate effectively with the study staff.
* Females must be using an acceptable method of contraception such as: abstinence, double barrier (condom, diaphragm, or cervical cap with spermicidal foam, gel, or cream), intrauterine device or hormonal contraception (oral, injectable, implantable, transdermal, or vaginal) used consecutively for at least 3 months prior to screening visit, vasectomized partner or use of implants for at least 6 months prior to screening visit; bilateral tubal ligation, hysterectomy, bilateral oophorectomy, or be postmenopausal status with amenorrhea (no menses) for at least 1 year prior to the screening visit.

Exclusion Criteria:

* Have a known sensitivity or allergy to any of the study products or their ingredients
* Have any medical condition or disease based on the professional judgement and experience of the principal investigator (PI) plus research industry standards that might affect or impact the administration of study products
* Lactating, pregnant or planning to become pregnant during the study
* History of drug or alcohol abuse in the 12 months prior to screening
* History of psychiatric illness requiring hospitalization in the 6 months prior to screening
* History of diabetes (Type I or II) or uncontrolled hypertension (either systolic BP >160 or diastolic BP >90)
* Participation in or use of a research IP within 30 days prior to screening (cannot have been in another study within 30 days of screening)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Cognition | 21 days
  Cognitive performance on the NIH Toolbox Cognition Battery and Joggle Psychomotor Vigilance Task. T scores (higher is better) will be reported.
Mood | 21 Days
  Self-reported Mood using the Mood and Physical Sensation Scale (higher scores reflect better mood)
Physical Performance | 21 Days
  Time to Exhaustion (TTE) Test - running on a treadmill with an increased incline every minute until perceived exhaustion is reached

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Tartar, Ph.D., Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kongkeaw C, Dilokthornsakul P, Thanarangsarit P, Limpeanchob N, Norman Scholfield C. Meta-analysis of randomized controlled trials on cognitive effects of Bacopa monnieri extract. J Ethnopharmacol. 2014;151(1):528-35. doi: 10.1016/j.jep.2013.11.008. Epub 2013 Nov 16. PMID 24252493
- [Background] Heaton RK, Akshoomoff N, Tulsky D, Mungas D, Weintraub S, Dikmen S, Beaumont J, Casaletto KB, Conway K, Slotkin J, Gershon R. Reliability and validity of composite scores from the NIH Toolbox Cognition Battery in adults. J Int Neuropsychol Soc. 2014 Jul;20(6):588-98. doi: 10.1017/S1355617714000241. Epub 2014 Jun 24. PMID 24960398
- [Background] Pickering C, Kiely J. What Should We Do About Habitual Caffeine Use in Athletes? Sports Med. 2019 Jun;49(6):833-842. doi: 10.1007/s40279-018-0980-7. PMID 30173351